CLINICAL TRIAL: NCT02808780
Title: Long-term Exposure Registry of Adult Patients With Moderate-to-Severe Ulcerative Colitis
Brief Title: An Observational Prospective Long-term Exposure Registry of Adult Patients With Moderate-to-Severe Ulcerative Colitis
Acronym: OPAL
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105891; CNTO148UCO4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-05-30; First posted 2016-06-22 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Simponi (Golimumab); Thiopurines; Lymphoma; Malignancies
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simponi-exposed cohort: Participants receiving Simponi at enrollment and are still receiving Simponi after participation in a therapeutic trial or participants scheduled to receive Simponi within 30 days after enrollment. Participants in this cohort may be receiving Simponi alone or in combination with thiopurines but must not be receiving other approved biologics or investigational agents at enrollment. Participants may have received other approved biologics or investigational agents prior to enrollment.
- Thiopurine cohort: Participants currently receiving thiopurines, having received at least 12 consecutive weeks of therapy prior to registry entry. Participants must not be receiving approved biologic agents, including Simponi, or investigational agents at enrollment. These patients may have received biologics other than Simponi or investigational agents prior to enrollment.

SUMMARY:
The purpose of this study is to describe the long-term safety risks in adult participants with moderate-to-severe ulcerative colitis who are treated with Simponi.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate-to-severe ulcerative colitis of at least 3 months' duration prior to enrollment, confirmed by endoscopy at any time in the past
* For enrollment into the Simponi-exposed cohort meets one of the following:

  1. The participant is currently receiving Simponi ,or
  2. The participant is continuing to receive Simponi after participation in an ulcerative colitis study, or
  3. The participant is scheduled to receive Simponi within 30 days after enrollment
* For Thiopurine cohort:

  1. The participant is currently receiving thiopurines, having received at least 12 consecutive weeks of therapy prior to registry entry
  2. Participant must not be receiving other approved biologic agents, including Simponi, or any investigational agents at enrollment
  3. Participant may have received biologics other than Simponi or investigational agents prior to enrollment

Exclusion Criteria:

* Participants who cannot be treated with Simponi or thiopurines
* Participants with a previous diagnosis of lymphoma or hematologic malignancy at any time prior to enrollment
* Participants currently receiving an investigational or biologic agent other than Simponi
* Participants with any condition for which, in the opinion of the investigator, participation in the registry would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate-to-severe ulcerative colitis for at least 3 months prior to enrollment will be observed
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Long-term Safety: Participants with Adverse Events of Interest (AEIs) and Serious Adverse Events (AEs) Including Malignancies, Pregnancies, and Non-serious Malignancies | 6 years
  Descriptive analysis of serious adverse events, adverse events of interest (including lymphoma & other malignancies), pregnancies, and non-serious malignancies in participants less than (<) 30 years of age will be reported.

SECONDARY OUTCOMES:
Clinical Disease Status as Assessed by Partial Mayo Score | 6 years
  The partial Mayo score, a validated tool used to assess disease status in participants with ulcerative colitis, will be utilized to assess clinical status in this registry. Information will be obtained using 3 of the individual components of the full Mayo score, including stool frequency, rectal bleeding, and PGA (Physician's Global Assessment). Each component score ranges from 0 (normal) to 3 (severe disease) and the score is the sum of those three categories. The total Partial Mayo Score will be calculated as the sum of the scores of all 3 components for each participant that ranges from 0-9.
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score | 6 years
  The SIBDQ is a disease-specific health-related quality of life (HRQoL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) patients by measuring physical, social and emotional status. The total score ranges from 10 (worst health) to 70 (best health).
EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L) Score | 6 years
  The EQ-5D-5L is a standardized non-disease specific instrument for describing and assessing health-related quality of life.This instrument evaluates 5 areas including mobility, ability for self-care, ability in usual activities, pain/discomfort and anxiety/depression.There also is a self-evaluated 100-point health assessment.
Work Productivity and Activity Impairment Questionnaire - Ulcerative Colitis (WPAI-UC) | 6 years
  The WPAI-UC is a validated instrument that measures the effect of ulcerative colitis (UC) symptoms on a patient's life (eg, diarrhea, loss of appetite, weight loss, abdominal pain, fever, joint pain, skin sores, rectal bleeding) and on his or her ability to work and perform regular activities.
Treatment Satisfaction Questionnaire for Medication (TSQM) Score | 6 years
  The TSQM is a 14-question instrument that gauges a patient's experience with his or her medication.The questionnaire was designed to evaluate the effectiveness, side effects, and convenience of the medication over a period of 2- to 3-weeks or since the last time it was taken.
Health Care Utilization: Evaluate the Number of Each Hospitalizations in Participants in Each Cohort | 6 years
  Number of hospitalizations in participants in each cohort will be reported.
Health Care Utilization: Evaluate the Reasons for Hospitalization in Participants in Each Cohort | 6 years
  Reasons for hospitalization in participants in each cohort will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (63):
- United States (16):
  - Murrieta, California
  - Rialto, California
  - Ventura, California
  - Coral Gables, Florida
  - Fort Myers, Florida
  - Lake Worth, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Tampa, Florida
  - Suwanee, Georgia
  - Chicago, Illinois
  - Sylvania, Ohio
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Lansdowne Town Center, Virginia
- Austria (3):
  - Salzburg
  - Sankt Poelten Noe
  - Vienna
- Canada (4):
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Oshawa, Ontario
  - Ottawa, Ontario
- Pilsen, Czechia
- France (9):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Grenoble
  - Montpellier
  - Nice
  - Pierre-Bénite
  - Saint-Priest-en-Jarez
  - Strasbourg
- Germany (11):
  - Berlin
  - Dessau Roblau
  - Halle
  - Hamburg
  - Heidelberg
  - Kiel
  - Leipzig
  - Ludwigshafen
  - Lyneburg
  - München
  - Saarbrücken
- Greece (4):
  - Athens
  - Heraklion
  - Ioannina
  - Thessaloniki
- South Korea (4):
  - Busan
  - Gyeonggi-do
  - Seongnam-si
  - Seoul
- Spain (11):
  - A Coruña
  - Barcelona
  - Córdoba
  - Fuenlabrada
  - Huelva
  - Madrid
  - Majadahonda
  - San Sebastián de los Reyes
  - Valencia
  - Vigo
  - Zaragoza